CLINICAL TRIAL: NCT03653117
Title: Transperineal Laser Ablation for Treatment of LUTS Due to Benign Prostatic Obstruction
Brief Title: Transperineal Laser Ablation for Treatment of Benign Prostatic Obstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Elesta S.R.L. (Industry)
Responsible Party: Principal Investigator, Prof.dr. H.P. Beerlage, Chairman of the Urology department, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018_149
Record Dates: First submitted 2018-08-22; First posted 2018-08-31 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Prostatic Hyperplasia, Benign
Keywords: Transperineal laser ablation; LUTS; BPO; Laser ablation
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Intervention Model Description: This study is a prospective, single centre, interventional pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TPLA (Experimental): TPLA procedure
  Interventions: Device: Transperineal laser ablation

INTERVENTIONS:
Device: Transperineal laser ablation — Minimal invasive coagulation of prostatic tissue by laser
  Other Names: Echolaser X4

SUMMARY:
Rationale: With age a large group of men experience lower urinary tract symptoms (LUTS) due to benign prostatic obstruction (BPO). Standard treatment is a transurethral resection of the prostate or laser vaporization. As these techniques enter the prostate via the urethra, are invasive and require general or spinal anaesthesia. Transperineal laser ablation (TPLA) is a minimal invasive procedure, that can be performed under local anaesthesia.

Objective: The primary objective of this study is to prove feasibility and safety of TPLA for LUTS due to BPO in healthy men.

Secondary objectives: The secondary objectives are to determine functional voiding, erectile outcomes and changes on imaging.

DETAILED DESCRIPTION:
This study is set up as a prospective, single centre, interventional pilot study.

Eligible patients are diagnosed with LUTS due to BPO at the outpatient clinic of the department of Urology at the Academic Medical Center (AMC) and have an indication for surgical treatment. The investigators aim to include 20 patients.

Eligible patients will be informed about this study by the urologist in the outpatient clinic. Information about the study will be provided both orally and in written form.

The TPLA procedure is performed with the Echolaser X4 system. The system uses a diode laser source that operates at the 1064nm wavelength. The maximum energy delivered is 10 watts per laser source. The system works with the concept of thermoablation, resulting in coagulative necrosis of tissue. Two to four fibers are introduced in the prostate under untrasound vision. Ablation will be performed with 3 watts power per fibre and a total of 1200 - 1800 J will be delivered per fibre in 400 - 600 s.

Follow-up will exist of four visits following surgery at 4 weeks, three, six and 12 months. The visits imply medical history, adverse event registration, physical examination (on indication) and uroflowmetry. Patient-reported outcome measures (PROMs) are used to measure functional outcomes. Used PROMs are the International Prostate Symptom Score (IPSS), International Index of Erectile Function 15 (IIEF-15), Visual Analogue Scale (VAS) and hematuria grading scale (HGS). In addition to this, imaging will exist of a contrast enhanced ultrasound (CEUS) at four weeks and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Male
* ≥ 40 years of age
* Peak urinary flow rate (Qmax): ≥ 5 mL/sec to ≤ 15 mL/sec, with a minimum voided volume of ≥ 125 mL, measured with uroflowmetry or urodynamic investigation
* Post-void residual (PVR): ≤ 250 mL
* Prostate volume: ≥ 30 and ≤ 120 cc, measured by transrectal ultrasound
* Urodynamic investigation proven bladder outlet obstruction
* Signed informed consent

Exclusion Criteria:

* Previous invasive prostate intervention (TURP, laser, ablation, etc.)
* History of prostate or bladder cancer
* Indwelling Foley catheter or clean intermittent catheterization (CIC)
* PSA of ≥ 3.0 ng/mL without negative biopsies
* Inability or unwillingness to tolerate temporary discontinuation of anticoagulation or anti-platelet therapy
* Other conditions / status

  * Active urinary tract infection / prostatitis
  * Macroscopic haematuria without a known contributing factor
  * Poor detrusor muscle function or other neurological disorder that would impact bladder function (eg, multiple sclerosis, Parkinson's disease, spinal cord injuries, (diabetic) polyneuropathy)
  * Concurrent malignancy except basal skin cancer
  * History of lower urinary tract surgery (eg, TURP, laser, urinary diversion, artificial urinary sphincter, penile prosthesis)
  * History of pelvic radiation therapy or radical pelvic surgery
  * History of bladder neck contracture and/or urethral strictures within the 5 years prior to the informed consent date
  * Bladder stones
  * Medical contraindication for undergoing TPLA surgery (eg, infection, coagulopathy, significant cardiac or other medical risk factors for surgery)
  * Diagnosed or suspected bleeding disorder

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
Incidence of technical successful TPLA treatments | 24 hours following TPLA treatment
  Number of technical successful performed TPLA treatments without failures related to the machine or procedure.
Incidence of TPLA treatment-emergent adverse events | 30 days following TPLA treatment
  Number of adverse events using the CTCAE v5.0. Procedural safety is shown when there are no adverse events of grade 3 or higher.

SECONDARY OUTCOMES:
Functional outcomes of TPLA | 12 months following TPLA treatment
  Functional outcomes of TPLA measured by uroflowmetry, expressed in change of Qmax.
Spontaneous voiding post TPLA | 24 hours following TPLA treatment
  The presence of spontaneous voiding following TPLA treatment
Erectile function | 12 months following TPLA treatment
  To evaluate erectile function after TPLA treatment, measured by the International Index of Erectile function 15 (IIEF-15) IIEF is a self-administered scale designed to assess erectile functioning: includes 15 questions on 5 relevant domains of male sexual function; Erectile function: Q1-5 Score range 0-5 + Q15 score range 1-5, total score 1-30, higher indicates better outcome; Orgasmic function: Q9-10 Score range 0-5, total score 0-10, higher indicates better outcome; Sexual desire: Q11-12 Score range 1-5, total score 2-10, higher indicates better outcome; Intercourse satisfaction: Q6-8 Score range 0-5, total score 0-15, higher indicates better outcome; Overall satisfaction: Q13-14 Score range 1-5, total score 2-10, higher indicates better outcome; All subscale are summed to combine them to a total IIEF-15 score.
Antegrade ejaculation | 12 months following TPLA treatment
  To evaluate antegrade ejaculation after TPLA treatment, measured by patient reporting.

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van Kollenburg RAA, van Riel LAMJG, Oddens JR, de Reijke TM, van Leeuwen TG, de Bruin DM. Contrast-enhanced Ultrasound Imaging Following Transperineal Laser Ablation for Lower Urinary Tract Symptoms. Urology. 2025 Apr;198:141-147. doi: 10.1016/j.urology.2024.11.043. Epub 2024 Nov 26. PMID 39603354